CLINICAL TRIAL: NCT03281746
Title: Effect of Prevention Education on Factors of Importance in Caries Formation in Pediatric Patients With Leukemia
Brief Title: Effect of Prevention Education in Caries Formation in Pediatric Patients With Leukemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-16-13019; NCI-2017-01354 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-09-07; First posted 2017-09-13 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Dental Care; Educational Status; Methods; Interviews as Topic; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (standard prevention education) (Active Comparator): Patients undergo dental examination at baseline and then receive standard prevention education at diagnosis discussing the effects of prolonged neutropenia on oral hygiene, importance of a regular oral hygiene regimen, and the long term clinical outcomes of oncologic patients. Patients also receive fliers with pictograms describing proper brushing, use of mouth wash, and common oral complications during therapy, as well as a bottle and prescription for chlorhexidine gluconate 0.12% rinse.
  Interventions: Procedure: Dental Procedure; Other: Educational Intervention (prevention education); Other: Interview; Other: Survey Administration
- Group II (standard and one-on-one education, consultation) (Experimental): Patients undergo dental examination and receive standard prevention education as in Group I. Patients also receive one-on-one prevention education and counseling with the physician and pediatric dental resident.
  Interventions: Procedure: Dental Procedure; Other: Educational Intervention (prevention education); Other: Interview; Other: Survey Administration; Other: Educational Intervention (one-on one education)

INTERVENTIONS:
Procedure: Dental Procedure — Undergo dental examination
Other: Educational Intervention (prevention education) — Receive prevention education
  Other Names: Education for Intervention; Intervention by Education
Other: Interview — Ancillary studies
Other: Survey Administration — Ancillary studies
Other: Educational Intervention (one-on one education) — Receive one-on-one education
  Other Names: Education for Intervention; Educational Intervention; Intervention by Education; Intervention through Education
  Arms: Group II (standard and one-on-one education, consultation)

SUMMARY:
This randomized pilot clinical trial studies how well preventive education works in decreasing caries formation in pediatric patients with leukemia. Prevention education may have an effect on factors important in causing cavities in pediatric patients with leukemia.

DETAILED DESCRIPTION:
Patients treated for leukemia at Virginia Commonwealth University Medical Center in the department of Pediatric Hematology and Oncology are currently receiving oral hygiene instruction at diagnosis. In this study, patients will be randomized into two groups at diagnosis: one receiving current prevention education and the other group receiving one-on-one prevention education and counseling with the physician and pediatric dental resident. Physician and pediatric dental resident will use motivational interviewing informed techniques during counseling. A caries risk assessment will be performed for each patient at diagnosis. Caries incidence, plaque scores, mutans streptococci levels, salivary flow rate, and salivary pH will be assessed at week one (diagnosis), week 16 or start of interim maintenance therapy whichever comes second, week 32 or beginning of maintenance therapy whichever is later for all patients enrolled in the study. Data will be collected through a clinical intraoral examination and salivary sample. Data collected will be used to assess the effect of increased prevention education on factors of importance in caries formation.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who have been recently diagnosed with leukemia
* Patients will also predictably be in primary or mixed dentition
* Patients of Virginia Commonwealth University Medical Center Pediatric Hematology Oncology Clinic

Exclusion Criteria:

* Full permanent dentition
* Primary language is not English
* Children in the custody of the state with no parent or legal guardian present to sign consent

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Change in caries assessed by CAMBRA risk assessment tool | Baseline up to 32 weeks
Change in salivary flow rate | Baseline up to 32 weeks
  Change in salivary flow rate will be measured utilizing pre-weighed cotton rolls. Patients will saturate as many cotton rolls as possible in one minute by chewing. Dose cups and cotton rolls will be weighed prior to and after data collection. The change in weight in grams will be converted to mL of saliva collected.
Change in salivary pH | Baseline up to 32 weeks
  Will be measured with litmus paper in the gingival sulcus of the tooth where plaque is collected for bacterial load testing.
Change in levels of mutans streptococci in buccal surface of most posterior maxillary right tooth | Baseline up to 32 weeks
  Samples will be plated on mitis salivarius and incubated. Mutans streptococci colonies will be counted after incubation.
Change in caries assessed by Merged International Caries Detection and Assessment System (ICDAS) | Baseline up to 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helou A Marieka, MD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States